CLINICAL TRIAL: NCT04711044
Title: Characterization of New Human Models of Non-histaminergic Itch and Their Interaction With the TRPM8 Receptor
Brief Title: Investigation of a New Human Model for Itch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Silvia Lo Vecchio, PhD, Assistant Professor, Aalborg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: N-20200005 (third sub-project)
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Itch
MeSH Terms: conditions — Pruritus | interventions — Papain; Histamine; Menthol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental)
  Interventions: Other: Papain; Other: Histamine; Other: Cowhage; Other: L-menthol

INTERVENTIONS:
Other: Papain — Papain will be applied using cowhage spicules inactivated by heat
Other: Histamine — To deliver histamine, standard allergy skin prick test (SPT) lancets are applied
Other: Cowhage — Cowhage spicules are 1-2 mm in length and have a diameter of 1-3 μm. The spicules are inserted by gently rubbing 30-35 spicules into a 1 cm diameter skin area.
Other: L-menthol — A 1 mL aliquot is dispensed onto a 2,5 × 2,5 cm cotton pad and placed on a 6 × 6 cm sheet of medical tape.

SUMMARY:
This third sub-project aims to evaluate the interaction between the TRPM8 receptor and pruritus by studying the anti-pruritic effect of TPRM8-agonist L-menthol on histaminergic and non-histaminergic itch induced using three different pruritogens: histamine, cowhage and papain.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* 18-60 years
* Speak and understand English

Exclusion Criteria:

* Pregnancy or lactation
* Drug addiction defined as any use of cannabis, opioids or other addictive drugs
* Previous or current history of neurological, dermatological, immunological musculoskeletal, cardiac disorder or mental illnesses that may affect the results (e.g. neuropathy, muscular pain in the upper extremities, etc.).
* Lack of ability to cooperate
* Current use of medications that may affect the trial such as antihistamines, antipsychotics and pain killers, as well as systemic or topical steroids.
* Skin diseases
* Moles, scars or tattoos in the area to be treated or tested.
* Hypersensitivity to papaya and mango fruit, cashew nuts, rubber latex
* Consumption of alcohol or painkillers 24 hours before the study days and between these
* Acute or chronic pain
* Participation in other trials within 1 week of study entry (4 weeks in the case of pharmaceutical trials)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-05 (Actual)

PRIMARY OUTCOMES:
Measuring itch intensity by computerized Visual Analog Scale Scoring | For 15 minutes
  We will ask the subjects to rate the sensation of itch on a 100 mm VAS scale ranging from 0 to 100 where 0 indicates "no itch" and 100 indicates "worst itch imaginable
Measuring pain intensity by computerized Visual Analog Scale Scoring | For 15 minutes
  We will ask the subjects to rate the sensation of pain on a 100 mm VAS scale ranging from 0 to 100 where 0 indicates "no pain" and 100 indicates "worst pain imaginable".
Superficial blood perfusion measurement | After 15 minutes
  Superficial blood perfusion is measured by a Speckle contrast imager
Measuring Alloknesis | 15 minutes
  Alloknesis is measured by using mildly pruritic, non-painful von Frey nylon filaments of a predetermined intensity (generally 5-30 milliNewton of force).

SECONDARY OUTCOMES:
Measurement of Cold Detection Thresholds (CDT) | 15 minutes
  The tests for thermal sensation will all be conducted using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device.
Measurement of Cold PainThresholds (CPT) | 15 minutes
  The tests for thermal sensation will all be conducted using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device.
Measurement of Heat Pain Thresholds (HPT) | 15 minutes
  The tests for thermal sensation will all be conducted using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device.
Measurement of Warm Detection Thresholds (WDT) | 15 minutes
  The tests for thermal sensation will all be conducted using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device.
Measurement of Pain to Supra-threshold Heat Stimuli | 15 minutes
  The tests for thermal sensation will all be conducted using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device.
Measurement of Mechanical Pain Thresholds (MPT) | 15 minutes
  This test is conducted using a pin-prick set.
Measurement of Mechanical Pain Sensitivity (MPS) | 15 minutes
  This test is conducted using a pin-prick set.
Touch Pleasantness (TP) | 15 minutes
  Pleasant touch sensation measured using a standardized sensory brush

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University, Aalborg, North Denmark, Denmark